CLINICAL TRIAL: NCT03499275
Title: MUscle STimulation in Advanced Idiopathic Pulmonary Fibrosis: a Randomised Placebo-controlled Trial
Brief Title: Muscle Stimulation in Advanced Idiopathic Pulmonary Fibrosis
Acronym: MUST-IPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Kings Clinical Trials Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 241055
Record Dates: First submitted 2018-04-11; First posted 2018-04-17 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Neuromuscular electrical stimulation
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: This is a study that comprises:
  * A parallel group, randomised placebo-controlled, assessor-blinded trial with participants randomised (1:1) to usual care (home based exercise programme) with either placebo or active NMES for six weeks, with a 12 week follow-up.
  * Qualitative interviews with participants and staff.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham NMES (Sham Comparator): Sham neuromuscular electrical stimulation plus home exercise programme and advice on breathlessness management
  Interventions: Device: Sham NMES; Other: Home exercise programme; Other: Breathlessness advice
- Active NMES (Experimental): Neuromuscular electrical stimulation plus home exercise programme and advice on breathlessness management
  Interventions: Device: Active NMES; Other: Home exercise programme; Other: Breathlessness advice

INTERVENTIONS:
Device: Active NMES — Neuromuscular electrical stimulation to the quadriceps muscle
  Arms: Active NMES
Device: Sham NMES — Sham neuromuscular electrical stimulation to the quadriceps muscle
  Arms: Sham NMES
Other: Home exercise programme — Home exercise programme. Both arms of the trial receive this intervention.
Other: Breathlessness advice — Breathlessness advice. Both arms of the trial receive this intervention.

SUMMARY:
The aims of this study are to determine whether neuromuscular stimulation (NMES) of the quadriceps muscle is acceptable to patients with Idiopathic Pulmonary Fibrosis (IPF) and staff and whether it can impact clinical and healthcare resource usage outcomes.

.

DETAILED DESCRIPTION:
Patients with IPF who consent to participate in the study will be allocated by chance to use 'active' or 'sham/placebo' NMES for six weeks. Patients will also complete a home exercise programme and receive advice on how to manage breathlessness. Clinical outcomes and trial flow after this six week programme and six weeks after patients have stopped using NMES will be assessed. After this point, healthcare resource use during the study period will be evaluated and interviews involving participants, their carers, and staff about their experiences of the study and using or delivering NMES will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF according to international standards.
* Severe respiratory disability / breathlessness (Medical Research Council dyspnoea score ≥3).
* Able to provide written informed consent.
* Declined or failed to complete a supervised centre-based pulmonary rehabilitation (PR) programme
* Quadriceps maximum voluntary contraction <80% predicted.

Exclusion Criteria:

* Cardiac pacemaker.
* Co-existing neurological condition.
* Change in medication or exacerbation requiring admission in preceding four weeks.
* Current regular exerciser (structured supervised training ≥3 times per week within last month).
* People who have completed PR in the previous six months.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | Six weeks
  Exercise capacity

SECONDARY OUTCOMES:
Quadriceps maximum voluntary contraction | Six weeks and twelve weeks
  Muscle strength
Rectus-femoris cross-sectional area | Six weeks and twelve weeks
  Muscle size
King's Brief Interstitial Lung Disease questionnaire | Six weeks and twelve weeks
  Measure of health-related quality of life that includes three domains (psychological, breathlessness and activities, chest symptoms) and a total score. The score range for each domain and the total score ranges from 0 to 100 with higher scores indicating better health-related quality of life.
Six minute walk test | Twelve weeks
  Exercise capacity

CONTACTS AND LOCATIONS:
Overall Officials: William DC Man, PhD, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, Harefield, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nolan CM, Patel S, Barker RE, Walsh JA, Polgar O, Maddocks M, George PM, Renzoni EA, Wells AU, Molyneaux PL, Kouranos V, Chua F, Maher TM, Man WD. Muscle stimulation in advanced idiopathic pulmonary fibrosis: a randomised placebo-controlled feasibility study. BMJ Open. 2021 Jun 2;11(6):e048808. doi: 10.1136/bmjopen-2021-048808. PMID 34083348